CLINICAL TRIAL: NCT05927532
Title: Argyle Fistula Cannula Pre-market, Prospective, Single Arm, Non-randomized, Interventional Study
Brief Title: Argyle Safety Fistula Cannula With Anti-reflux Valve Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT19046
Record Dates: First submitted 2023-01-19; First posted 2023-07-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Argyle Fistula Cannula Subjects (Experimental): All subjects enrolled in the study and treated with the Argyle Safety Fistula Cannula with Anti-reflux Valve
  Interventions: Device: Argyle Safety Fistula Cannula with Anti-Reflux Valve

INTERVENTIONS:
Device: Argyle Safety Fistula Cannula with Anti-Reflux Valve — The Argyle Safety Fistula Cannula with Anti-reflux Valve will be used 3x a week for 12 weeks in subjects with an arteriovenous fistulae (AVF) fistula

SUMMARY:
The purpose of the investigation is to confirm the safety and performance of the Argyle™ Safety Fistula Cannula with Anti-reflux Valve for hemodialysis treatment.

DETAILED DESCRIPTION:
The study will be performed at up to 5 US hemodialysis clinics.

Qualified patients who choose to participate and sign informed consent will be enrolled in the study. The investigational sites chosen to participate in this study will be trained on the insertion procedure using plastic fistula cannulas according to established curriculum. A combination of didactic training followed by insertion using a cannulation arm will be conducted. Cannulation on consented subjects will begin after the inserter demonstrates proficiency on the cannulation arm. Proficiency definitions are outlined in the protocol. After two supervised (by Medtronic and/or dedicated, trained super user) successful cannulations on consented subjects, the clinician will be permitted to cannulate without supervision.

Data supporting the primary, secondary, and exploratory objectives will be captured following thirty-six (36) hemodialysis sessions for each enrolled subject.

Cannulations will be performed by a minimum of five different clinicians at up to 5 dialysis clinic sites.

The investigational sites chosen to participate in this study will be trained on the insertion procedure using plastic fistula cannulas for a pre-determined period and according to established curriculum. A combination of didactic training followed by insertion using a cannulation arm will be conducted. After two supervised (by Medtronic and/or dedicated, trained super user) successful cannulations on consented subjects, the clinician will be permitted to cannulate without supervision and the data collection for the primary and secondary objectives will begin. Hemodialysis sessions will be performed, according to the investigator's prescription, throughout the duration of the study. Dialysis adequacy will be verified at baseline and during the mid-week session on weeks 1, 3, 6 and 12. Other than the blood sampling, there are no study-specific procedures, other than cannulation with the Argyle™ Safety Fistula Cannula with Anti-Reflux Valve, that will be required.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is aged 18 years or older who signed informed consent
* Subject is undergoing in-center hemodialysis
* Subject has an arteriovenous fistulae (AVF) fistula that was determined to be mature by standard clinical definition

Exclusion Criteria:

* Subject is enrolled in another study that could confound the results of this study, without documented pre-approval
* Subject with an existing arteriovenous graft
* Subjects with known allergies to plastics
* Subjects who are unable to read or respond to the questionnaire about satisfaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Successful Hemodialysis Sessions | through study completion, an average of 1 year
  The primary objective is the percentage of successful hemodialysis sessions using the Argyle™ Safety Fistula Cannula with Anti-reflux Valve.

SECONDARY OUTCOMES:
Successful Cannulations | through study completion, an average of 1 year
  Report the percentage of successful cannulations to achieve successful cannulation in each subject
Cannulation Locations with securement details | through study completion, an average of 1 year
  Characterize cannulation locations and details on the securement of the cannulas after taping during the hemodialysis session by evaluating the staff-reported insertion sites captured on the Dialysis Session case report form
Access-related complications requiring procedural intervention | through study completion, an average of 1 year
  Quantify the number of subjects who had a procedure to correct access-related complications
Compare prescribed blood flow rates | through study completion, an average of 1 year
  Compare prescribed blood flow rates with plastic fistula cannula to average blood flow achieved
Dialysis adequacy | through study completion, an average of 1 year
  Compare baseline dialysis adequacy (e.g., spKt/V and urea reduction ratio (URR) to measure collected at 1, 3, 6 and 12 weeks). The average spKt/V and URR will be compared to measurements reported at basline using steel needles. A repeated measures approach will be utilized to compare baseline to follow-up dialysis adequacy measurements.
Cannulator Satisfaction Questionnaire | through study completion, an average of 1 year
  Assess inserter satisfaction (survey), i.e., ability to access deep fistulas, insertion locations, securement technique, ability to determine proper placement without the usual pulsing flashback seen with traditional needles. Mean satisfaction score (and associated 95% confidence intervals) prior to first use and following final cannulation will be reported.
Subject Satisfaction Questionnaire | through study completion, an average of 1 year
  Characterize subject satisfaction using standardized survey to assess insertion pain
Impact of delay between training and use of device | through study completion, an average of 1 year
  Evaluate any impact of delay between training and use of the subject devices, or time elapsed between cases for each clinician and successful and unsuccessful cannulations. The proportion of successful and unsuccessful cannulations will be predicted with clinician and time between training and cannulation attempt using logistic regression. Statistical significance of the covariate "time between training and cannulation attempt" will be reported.

OTHER OUTCOMES:
Summary of Needle Stick Injury within past 6 months from start of study by investigational site | in the past 6 months from the start of the study
  Summarize any reported needle stick injury reports in the past 6 months from the start of the study, as permitted by the investigational site
Time to successful cannulation | During procedure
  Report the time required to achieve successful cannulation

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - DaVita Hartford, Hartford, Connecticut
  - DaVita Columbus, Columbus, Georgia
  - DaVita Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No